CLINICAL TRIAL: NCT05803005
Title: Evaluation of Some Inflammatory Markers in Autism Spectrum Disorders
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Ghada Mohamed Ali, assiut, Assiut University
Other Study IDs: inflammatory markers in autism
Record Dates: First submitted 2023-03-26; First posted 2023-04-07 (Actual); Last update posted 2023-04-07 (Actual); Status verified 2023-03

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- children with autism spectrum disorder: : 50 patients aged 3_18 years, equally sex distributed, who visit pediatric neurology outpatients clinic with autistic disorder at assiut university hospital will enrolled in this study and 50 controls . (According to DSM IV and ADT-R)
  Interventions: Other: inflammatory marker in autism spectrum disorder

INTERVENTIONS:
Other: inflammatory marker in autism spectrum disorder — Evaluate some Inflammatory markers [IL-6, IL-8, TNF_alpha] in children with autism spectrum disorder

SUMMARY:
Evaluate some Inflammatory markers [IL-6, IL-8, TNF_alpha] in children with autism spectrum disorder

DETAILED DESCRIPTION:
several studies have suggested a correlation between ASD and abnormal immune activation (9) For instance, there is a high incidence of autistic subjects in families with other autoimmune disorders such as celiac disease and rheumatoid arthritis, suggesting a potential role for immune dysfunction in the pathophysiology of ASD High levels of IL-6 in the brain could determine alterations of synapse formation, dendritic spine development, and neuronal circuit balance [13], while in plasma they have been associated with increased stereotypical behaviors and with regressive forms of ASD

ELIGIBILITY:
Inclusion Criteria:

* 50 patients aged 3_18 years, equally sex distributed, who visit pediatric neurology outpatients clinic with autistic disorder at assiut university hospital will enrolled in this study and 50 controls . (According to DSM IV and ADT-R)

Exclusion Criteria:

* : Asperger syndrome, pervasive developmental disorder not otherwise specified (PDD-NOS), chronic seizures and recent infection and patients with congenital anomalies

Ages: 3 Years to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: : 50 patients aged 3_18 years, equally sex distributed, who visit pediatric neurology outpatients clinic with autistic disorder at assiut university hospital will enrolled in this study and 50 controls . (According to DSM IV and ADT-R)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
inflammatory marker in autism | baseline
  Evaluate some Inflammatory markers [IL-6, IL-8, TNF_alpha] in children with autism spectrum disorder

CONTACTS AND LOCATIONS:
Overall Officials: gehan kamal, prof., Study Director — assiut universtiy

IPD SHARING:
Plan to Share IPD: No